CLINICAL TRIAL: NCT01735409
Title: A Single Center Phase IIa Study of Nanoparticle Albumin-bound Paclitaxel in Combination With Cisplatin in Advanced Nasopharyngeal Carcinoma
Brief Title: Dose-finding Study of Abraxane in Combination With Cisplatin to Treat Advanced Nasopharyngeal Carcinoma
Acronym: ABX-DDP-Dose
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, Professor, Sun Yat-sen University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABXDDP20101224
Record Dates: First submitted 2012-11-22; First posted 2012-11-28 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Nasopharyngeal Neoplasms
Keywords: Advanced Nasopharyngeal Carcinoma; Abraxane; Cisplatin; Dose
MeSH Terms: conditions — Nasopharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1-day regimen (Experimental): ABX 260 mg/m2 day 1 + DDP 75mg/m2 day 1
  Interventions: Drug: ABX + DDP
- 2-day regimen (Experimental): ABX 140 mg/m2 day 1,8 + DDP 75mg/m2 day 1
  Interventions: Drug: ABX + DDP
- 3-day regimen (Experimental): ABX 100 mg/m2 day 1,8,15 + DDP 75mg/m2 day 1
  Interventions: Drug: ABX + DDP

INTERVENTIONS:
Drug: ABX + DDP — ABX 260 mg/m2 day 1 + DDP 75mg/m2 day 1
  Arms: 1-day regimen
Drug: ABX + DDP — ABX 140 mg/m2 day 1,8 + DDP 75mg/m2 day 1
  Arms: 2-day regimen
Drug: ABX + DDP — ABX 100 mg/m2 day 1,8,15 + DDP 75mg/m2 day 1
  Arms: 3-day regimen

SUMMARY:
This is a single center, non-randomized phase IIa study to determine the tolerance and safety of Abraxane (ABX) in combination with cisplatin (DDP) in patients with advanced nasopharyngeal carcinoma (NPC). Patients in whom the standard therapy had failed or had been infeasible will be eligible.The safety and efficacy will be evaluated according to NCI-CTCAE V4.0 and RECIST 1.1 respectively.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) is most commonly seen in Southeast Asia, especially in southern and southeastern China, where the incidence rate has been documented between 10 and 150 cases per 100,000 population per year. For advanced or metastatic NPC, chemotherapy remain the mainstay of treatment. The 130-nm albumin-bound formulation of paclitaxel ([Abraxane, ABX ];Celgene,Summit,NJ) is a promising new agent with more efficient entry to the tumor microenvironment via caveolae-mediated transcytosis and preferential uptake by cancer cells. Superior activity of ABX-based regimens without the necessity for antianaphylactic pretreatments been shown in various solid tumors compared with the traditional solvent-based paclitaxel-based ones. However, the safety and efficacy of combination of ABX and cisplatin (DDP) has not been determined in patients with advanced NPC. In this single center, non-randomized phase IIa study, investigators seek to determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of ABX-DDP, and perform an exploratory study of its efficacy as measured by tumor response.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven NPC diagnosis
* Patients who failed the prior standard treatment or were intolerant of standard treatment
* Elder than 18 years old
* Performance status 0-2
* Patients previously treated with chemotherapy (those having received paclitaxel-based regimen were not excluded)
* Subjects with at least one measurable lesion (Tumor lesions that are situated in a previously irradiated area could not be considered measurable).
* Life expectancy over twelve weeks
* Neutrophil > 1.5X10^9/L, PLT > 100X10^9/L, Hb ≥ 90 g／l, with normal hepatic function(AST, ALT < 2.5 x upper limit of normal , and bilirubin < 1.0 x upper limit of normal), with normal renal function (creatinine < 1.5 x upper limit of normal or creatinine clearance ≥ 60ml/min as calculated by the Cockcroft - Gault formula. )
* Urine pregnancy test (-) within 1 weeks before enrollment or being able to take effective contraceptive measures during the medication and six months after completion of the trial for fertile women.
* Being able to provide paraffin blocks or 5-7 slides of biopsy tumor tissues.
* Amenable to regular follow-up and to comply with trial requirements.
* Signed and dated informed consent before the start of specific protocol procedures

Exclusion Criteria:

* History of allergy to paclitaxel or docetaxel
* Patient with central nervous system metastasis
* Patient refusing participation or signing informed consent
* Active clinically serious infections with an anticipated antibiotics treatment for more than 4 weeks
* Patient with life threatening medical condition such as congestive heart failure, symptomatic coronary artery disease or heart block
* Myocardial infarction that occurred within 3 months before enrollment
* Had received chemotherapy, radiotherapy or other anti-cancer therapies within 3 weeks before enrollment
* With a pre-existing peripheral neuropathy (National Cancer Institute Common Toxicity Criteria for Adverse Events [NCI CTC] grade ≥ 2)
* Previously received post-2nd line anti-cancer therapy
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors[Ta, Tis & T1] or any cancer curatively treated > 3 years prior to study entry.
* History of immunodeficiency , including HIV testing positive or suffering from other acquired and congenital immunodeficiency disease, or the history of organ transplants;
* Patients receiving prior abraxane treatment during pregnancy or lactation period
* Fertile women who failed to or are reluctant to take contraceptive measures or pregnancy test
* Men or his companion who are reluctant to take effective contraceptive measures during the medication and six months after completion of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-03 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 24 months

SECONDARY OUTCOMES:
Progression free survival (PFS) | 24 months
Number of Participants with Adverse Events | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Huang Y, Liang W, Yang Y, Zhao L, Zhao H, Wu X, Zhao Y, Zhang Y, Zhang L. Phase I/II dose-finding study of nanoparticle albumin-bound paclitaxel (nab(R)-Paclitaxel) plus Cisplatin as Treatment for Metastatic Nasopharyngeal Carcinoma. BMC Cancer. 2016 Jul 13;16:464. doi: 10.1186/s12885-016-2517-5. PMID 27411683